CLINICAL TRIAL: NCT01639846
Title: A Single-Center, Double-Masked, Randomized, Vehicle Controlled Evaluation of the Onset and Duration of Action of RX-10045 Ophthalmic Solution, 0.09% Compared to Vehicle in the Conjunctival Allergen Challenge (CAC) Model of Allergic Conjunctivitis
Brief Title: Evaluation of the Onset and Duration of Action of RX-10045 in Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: C.T. Development America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTD1202
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — isopropyl 5,12-hydroxypentadeca-8,10-dien-6,14-diynoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- RX-10045 active arm (Experimental): RX-10045 Ophthalmic Solution, 0.09%
  Interventions: Drug: RX-10045
- Vehicle for RX-10045 arm (Placebo Comparator): Vehicle of RX-10045 Ophthalmic Solution
  Interventions: Drug: Vehicle for RX-10045 arm

INTERVENTIONS:
Drug: RX-10045 — RX-10045 Ophthalmic Solution, 0.09% At Visits 3A and 4, a trained study technician will instill one drop of the assigned, masked study treatment, into each eye.
  Arms: RX-10045 active arm
Drug: Vehicle for RX-10045 arm — Vehicle of RX-10045 Ophthalmic Solution At Visits 3A and 4, a trained study technician will instill one drop of the assigned, masked study treatment, into each eye.
  Arms: Vehicle for RX-10045 arm

SUMMARY:
To purpose of this study is to establish the efficacy and safety of RX-10045 ophthalmic solution in alleviating the signs and symptoms of allergic conjunctivitis

DETAILED DESCRIPTION:
Allergies are relatively common among the general population. Ocular signs and symptoms include itching, discomfort, redness, chemosis, tearing, and eyelid swelling. Allergic reactions can vary from a mild, self-limiting disease, to a debilitating condition that significantly impairs the quality of life of allergen-sensitive individuals.

Currently approved treatments for ocular allergy reduce the signs and symptoms of the early phase reaction; however, evidence suggests that many patients suffer from the persistent late phase reaction. Manifestations of the late phase reaction occur 6 to 24 hours after allergen exposure and are characterized by an influx of acute inflammatory cells into the conjunctivae. Administration of anti-inflammatory agents decreases allergy signs and symptoms in both the early and late phase reactions.

RX-10045 has been shown to be efficacious in multiple pre-clinical dry eye disease models and in a pre-clinical model of allergic conjunctivitis. The objective of this clinical study is to assess the safety and efficacy of RX-10045 ophthalmic solution for the treatment of the signs and symptoms of allergic conjunctivitis induced in the Conjunctival Allergen Challenge Model of allergic conjunctivitis at 15 minutes and 8 hours after medication instillation. It is anticipated that RX-10045 has therapeutic potential for the treatment of allergic conjunctivitis and an acceptable risk-benefit profile.

ELIGIBILITY:
Inclusion Criteria:

Subjects MUST:

1. Have a positive history of ocular allergies
2. Have a positive bilateral conjunctival allergen challenge (CAC) reaction

Exclusion Criteria:

Subjects MUST NOT:

1. Have known contraindications or sensitivities to study medication or its components
2. Have any ocular condition that, in the opinion of the investigator, could affect the subject's safety or trial parameters
3. Use a disallowed medication during the period indicated prior to the enrollment or during the study
4. Be a female who is currently pregnant, planning a pregnancy, lactating, or not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Ocular itching | Baseline to day 14
  Ocular itching at defined timepoints up to 2 weeks
Conjunctival redness | Baseline to day 14
  Conjunctival redness evaluated by the investigator at defined timepoints up to 2 weeks

SECONDARY OUTCOMES:
Ciliary and episcleral redness | Baseline to day 14
  Ciliary and episcleral redness evaluated by the investigator at defined timepoints up to 2 weeks
Chemosis | Baseline to day 14
  Chemosis evaluated by the investigator at defined timepoints up to 2 weeks
Eyelid swelling | Baseline to day 14
  Eyelid swelling evaluated by the subject at defined timepoints up to 2 weeks
Tearing | Baseline to day 14
  Tearing evaluated by the subject at defined timepoints up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States